CLINICAL TRIAL: NCT05102578
Title: Understanding Persistent Pain: A Feasibility Study for the Use of a Digital Decision Aid Tool for Persistent Pain in a Pharmacy Setting
Brief Title: Understanding Persistent Pain Using a Decision Aid Tool in a Scottish Pharmacy Setting.
Acronym: UPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: Pharmacy Research UK (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2021UA003E-281537
Record Dates: First submitted 2021-06-10; First posted 2021-11-01 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2022-07

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Care (No Intervention): Usual care. Consultation with pharmacist with no decision aid tool.
- Digital Decision Aid Tool (Experimental): Consultation with pharmacist using the digital decision aid tool.
  Interventions: Behavioral: Digital Decision Aid Tool

INTERVENTIONS:
Behavioral: Digital Decision Aid Tool — The digital DAT will ask people about their current pain levels, medications and physical activity. Following this, it will include a Discrete Choice Experiment (DCE)-like component with a series of questions that ask users to choose between different pain management packages. Similar to a standard DCE, packages (or plans) are described by attributes and levels, which include broad categories of guideline-based pain management strategies routinely available in clinical practice. The descriptors used for the attributes and levels were informed by a previous qualitative research study and based on therapeutic options that are helpful and important to people with persistent pain .
  Arms: Digital Decision Aid Tool

SUMMARY:
Persistent pain describes long term pain that is present nearly every day. It is common and affects millions of people in the United Kingdom. The investigators want to explore people's experience of living with persistent pain and investigate how pharmacists can help people manage their pain. For this, the investigators will be testing a digital Decision Aid Tool (DAT) that includes a pain and lifestyle assessment as part of a pain consultation.

DETAILED DESCRIPTION:
The study design is a randomised feasibility study. Patient participants will take part in a pain consultation with a pharmacist to discuss pain management in a shared decision making (SDM) process. The unit of randomisation will be the patient participant. Thus, pharmacists will randomise patients to one of two groups: an intervention group who will receive a digital DAT for self-completion as part of the consultation and a control group which not use the digital DAT.

How the study will be implemented will be dependent on research restrictions due to the COVID-19 pandemic. If restrictions on research are in place, all study activities will be done remotely. If research restrictions are lifted the investigators will offer both remote and in person activities, depending on the participants preference.

Registered pharmacists in National Health Service (NHS) Grampian (see Section 5.1.) will be invited to take part in the study. As part of the assessment of feasibility for a future randomised control trial (RCT), a mixture of community and General Practitioner (GP)-surgery based pharmacists will be recruited. Recruited pharmacists will identify and invite patients living with persistent pain to a pain consultation. Pharmacists and patients will discuss current lifestyle and pain history, after which the pharmacist will recommend pain management plans that follow a person centred care (PCC) approach. Patients in the intervention group will receive the digital DAT - named UPP (Understanding Persistent Pain) - for self-completion with the help of the pharmacist. The DAT will generate a personalised report on the patient's preferences that can be used to discuss different PCC management plans. Management plans will be based on strategies routinely available in clinical practice4.

Heterogeneity in pharmacist-led pain consultations means that consultations are likely to differ across pharmacists. This study will allow the researchers to characterise different types of pharmacist-led pain consultations for a future larger study. As such, having a standardised control consultation falls beyond the scope of this feasibility study. Similarly, heterogeneity in current practice will cause agreed plans to differ across pharmacists and patients. These will also depend on the prescribing qualifications of the pharmacist.

The patient's GP will be informed of the person's participation and, in some cases, the recommendations/findings of the consultation. Where a prescription only medicine is deemed beneficial, pharmacists who are qualified independent prescribers will recommend this directly. Pharmacists without this qualification will, with the agreement of the patient, suggest to patients that they should book an appointment with the GP and send a referral letter to the GP with the recommendation for the prescription only medicine. Follow up consultations with the pharmacist will be arranged according to each pharmacist's current practice.

Parallel to the study, a testing event with patients living with persistent pain will be organised. Participants will be recruited using posters in GP Practices and using local patient networks. Participants will attend a half day event where they will get to use the digital DAT with the research team and provide feedback. Informed consent will be taken by the research team prior to the start of the event.

ELIGIBILITY:
Inclusion Criteria:

* Above 18 years old.
* Suffer from non-malignant persistent pain (defined as pain lasting for more than three months).
* Managed entirely within a primary care setting.

Exclusion Criteria:

* Not fluent in the English language.
* Have concomitant severe mental health problems or terminal illness.
* Suffer from pain caused by cancer or other malignancy.
* Not able to give informed consent (e.g. because of mental state)
* Takes part in another research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Pain assessed using the Chronic Pain Grade | 6 weeks
  Self-administered questionnaire that records subscale scores for pain intensity and disability are combined to calculate a chronic pain grade that enables classification of chronic pain patients.
EuroQol's 5D-5L | 6 weeks
  Self-administered questionnaire that records state and quality of life using EuroQol's five dimensions and 5 levels.
Personal Well-being Scale | 6 weeks
  Self-administered questionnaire that records personal wellbeing using the UK's Office of National Statistics (ONS) Measuring Subjective Well-being for Public Policy.

CONTACTS AND LOCATIONS:
Overall Officials: Mandy Prof Ryan, Principal Investigator — HERU Director
Locations (2):
- United Kingdom (2):
  - NHS Grampian, Aberdeen
  - University of Aberdeen, Aberdeen

IPD SHARING:
Plan to Share IPD: Yes
Any data shared with other researchers will be anonymised.
Supporting Information: Study Protocol, ICF
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Individual participant data (after de-identification) that underlie the results of this study will be available upon reasonable requests to investigators whose proposed used of data has been approved by an independent review committee identified for this purpose.
URL: https://www.abdn.ac.uk/achds/index.php

REFERENCES:
- [Derived] Loria-Rebolledo LE, Ryan M, Bond C, Porteous T, Murchie P, Adam R. Using a discrete choice experiment to develop a decision aid tool to inform the management of persistent pain in pharmacy: a protocol for a randomised feasibility study. BMJ Open. 2022 Sep 22;12(9):e066379. doi: 10.1136/bmjopen-2022-066379. PMID 36137622